CLINICAL TRIAL: NCT04219176
Title: Spectral Optical Coherence Tomography Findings in Patients With Ocular Toxoplasmosis : a Retrospective Study
Brief Title: Spectral Optical Coherence Tomography Findings in Patients With Ocular Toxoplasmosis
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, clinical professor, Université de Sousse
Other Study IDs: U23454
Record Dates: First submitted 2019-12-28; First posted 2020-01-06 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ocular Toxoplasmosis
Keywords: Spectral optical coherence tomography; Ocular toxoplasmosis; Uveitis
MeSH Terms: conditions — Toxoplasmosis, Ocular; Uveitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spectral optical coherence tomography — Swept-source optical coherence tomography (SS-OCT) is the latest milestone in retinal and choroidal imaging. Because its wavelength of 1050 nm, which is superior to the 840 nm of spectral domain optical coherence tomography (SD-OCT), it is able to overcome ocular opacities such as cataracts and vitritis, wich allows retinal and choroidal visualization of eyes whose fundus is not clearly visible. Consequently , SS-OCT allows visualization of the retinal and choroidal vascular networks, even in eyes with medium opacity

SUMMARY:
Ocular toxoplasmosis is the most common cause of infectious uveitis worldwide. The diagnosis of ocular toxoplasmosis is primarily clinical when it is a typical presentation .With an atypical presentation in the fundus, parasitological diagnosis is a decisive contribution, as well as multimodal imaging. We investigate on vitreal, retinal, and choroidal morphologic changes in active and scarred toxoplasmosis lesions using swept source optical coherence tomography.

DETAILED DESCRIPTION:
A retrospective analysis of patients diagnosed with ocular toxoplasmosis was conducted. The patients were examined at ophthalmology service of Farhat Hached Hospital in Sousse Tunisia between January 2002 and December 2017. Complete ophthalmologic examination and OCT were done at the initial visit and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized for ocular toxoplasmosis.

Exclusion Criteria:

* patients with non active ocular toxoplasmosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nine eyes of nine patients consecutively diagnosed with ocular toxoplasmosis were included in this retrospective study. The patients were examined at ophthalmology service of Farhat Hached Hospital in Sousse Tunisia between January 2002 and December 2017
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2002-01-23 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
number of prticipant affected with ocular toxoplasmosis | up to one year
  patient diagnosed having ocular toxoplasmosis

IPD SHARING:
Plan to Share IPD: No